CLINICAL TRIAL: NCT03569462
Title: mHealth and HIV Self-testing for High-risk Men in China
Brief Title: mHealth and HIV Self-testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Anhui Medical University (Other); University of Arkansas (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Don Operario, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH106349 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2018-06

CONDITIONS: Mobile Health Intervention to Promote HIV Self-testing
Keywords: HIV self-testing; Mobile Health; Men who have sex with men; China
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Intervention Model Description: Intervention involves demonstration of HIV self-testing and access to a mobile health application to promote HIV self-testing and HIV behavioral risk reduction
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile "WeChat" intervention (Experimental): Participants will watch a demonstration of HIV self-testing, receive HIV self-testing kits, and receive access to a mobile health application that delivers content to promote HIV-self testing and reduce HIV-related risk behavior.
  Interventions: Behavioral: Mobile "WeChat" intervention
- Control condition (Active Comparator): Participants will watch a demonstration of HIV self-testing and receive HIV self-testing kits.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Mobile "WeChat" intervention — Participants watch a demonstration of HIV self-testing, receive HIV self-testing kits, and receive access to a mobile application that delivers content to promote HIV self-testing and reduce HIV risk behavior
  Arms: Mobile "WeChat" intervention
Behavioral: Control condition — Participants watch a demonstration of HIV self-testing and receive HIV self-testing kits.
  Arms: Control condition

SUMMARY:
The investigators will pilot test an intervention to use a mobile application ("app") to improve HIV self-testing (HST) with high-risk men in China. Sixty participants will be randomly assigned to an intervention group - which involves access to a mobile app-based HIV testing health promotion and risk reduction program - versus control. Participants will be evaluated at baseline and at 6-month follow up with respect to HST and changes in sexual risk behaviors.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) have emerged as one of the fastest growing HIV risk populations in China, the world's most populous country. Studies in China report that MSM have low rates of HIV testing, low use of HIV prevention services, and high levels of unprotected sex with both male and female partners. Stigma presents one of the critical barriers to engaging MSM in HIV testing and prevention interventions, as many MSM in China avoid health service facilities that require face-to-face disclosure of their same-sex behaviors. Because HIV testing is a crucial opportunity for HIV prevention and represents the first step on the continuum of care, efforts to improve rates of HIV testing among MSM in China can contribute to reduced risk for HIV transmission and enhanced public health outcomes in this population.

For high-risk MSM in China, HIV self-testing (HST) offers a compelling strategy for achieving higher levels of HIV testing, due to the removal of barriers associated with traditional forms of in-person, clinic-based HIV testing. HST allows individuals to self-administer the HIV rapid diagnostic test in a private setting, which can detect for the presence of HIV-1/2 antibodies. The overarching goal of this research investigation is to improve the implementation science of HIV self-testing (HST) as a public health strategy to increase HIV testing among populations with low testing rates.

The investigators propose using a mHealth approach to support the implementation of HST. Specifically, the investigators hypothesize that incorporating mobile application- or "app"-based behavioral risk reduction messages with HST can preserve the privacy and comfort associated with self-administered testing, while also allowing for individuals to receive timely information and motivational cues to take the crucial next steps following their HST results - i.e., to test repeatedly, to reduce their behavioral risks for HIV transmission, and to seek appropriate referral services as needed.

This research will examine the acceptability and preliminary effects of HST linked with app-based behavioral risk reduction messages in a sample of high-risk MSM in China. In this pilot study, the investigators will test the primary hypothesis that the combination of HST plus mobile app-based risk reduction messaging compared to HST alone will increase HST re-testing and reduce sexual risk behavior in the next 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Biological male
* Unprotected anal sex during the past 6 months
* Current resident in Hefei (city), China
* HIV-negative or HIV-status unknown
* Possess a mobile "smart" phone
* Not planning to relocate from study location

Exclusion Criteria:

* HIV positive at enrollment
* Self-report coercion to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
HIV self-testing, picture | 6 months
  Picture of HIV self-test result submitted via mobile app
HIV self-testing, self-reported | 6 months
  Self-reported use of HIV self-test kit
HIV risk behavior | 6 months
  Condomless sex acts

CONTACTS AND LOCATIONS:
Overall Officials: Don Operario, PhD, Principal Investigator — Brown University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han L, Bien CH, Wei C, Muessig KE, Yang M, Liu F, Yang L, Meng G, Emch ME, Tucker JD. HIV self-testing among online MSM in China: implications for expanding HIV testing among key populations. J Acquir Immune Defic Syndr. 2014 Oct 1;67(2):216-21. doi: 10.1097/QAI.0000000000000278. PMID 24991972
- [Background] Tao J, Li MY, Qian HZ, Wang LJ, Zhang Z, Ding HF, Ji YC, Li DL, Xiao D, Hazlitt M, Vermund SH, Xiu X, Bao Y. Home-based HIV testing for men who have sex with men in China: a novel community-based partnership to complement government programs. PLoS One. 2014 Jul 22;9(7):e102812. doi: 10.1371/journal.pone.0102812. eCollection 2014. PMID 25051160
- [Background] Zhang C, Li X, Brecht ML, Koniak-Griffin D. Can self-testing increase HIV testing among men who have sex with men: A systematic review and meta-analysis. PLoS One. 2017 Nov 30;12(11):e0188890. doi: 10.1371/journal.pone.0188890. eCollection 2017. PMID 29190791